CLINICAL TRIAL: NCT01024426
Title: Evaluating the Impact of Enhanced Health Facility-based Care for Malaria and Febrile Illnesses in Children in Tororo, Uganda
Brief Title: Impact of Enhanced Health Facility Care in Uganda
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uganda Malaria Surveillance Project (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); University of California, San Francisco (Other); Infectious Diseases Research Collaboration, Uganda (Other)
Responsible Party: Principal Investigator, Sarah Staedke, Principal Investigator, Uganda Malaria Surveillance Project
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ITGBVG01
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Malaria
Keywords: Uganda; malaria; enhanced health facility-based care; febrile illnesses; health services
MeSH Terms: conditions — Malaria | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Health Facility intervention (Experimental): In the clusters randomized to enhanced health facility-based care, the intervention is designed to address these barriers and will focus on three components: (1) training in-charges in health center management, (2) providing training to health workers in fever case management and patient-centered services, and (3) ensuring adequate supplies of artemether-lumefantrine and RDTs.
  Interventions: Procedure: Enhanced health facility-based care
- Standard of care (Other): In the clusters randomized to standard care, standard care will include services typically provided by government-run facilities; we will not provide any additional support to these facilities. Health care will be provided to patients attending these facilities according to the usual standards; in-charges will continue to manage the facilities using their standard approach, no additional training will be provided to the health workers stationed at these facilities; and no support for staffing or supplies will be provided beyond what is supplied by the district and MoH.
  Interventions: Other: Standard care

INTERVENTIONS:
Procedure: Enhanced health facility-based care — The intervention is designed to address barriers to delivering quality care at health centers and will focus on three components: (1) training in-charges in health center management, (2) providing training to health workers in fever case management and patient-centered services, and (3) ensuring adequate supplies of artemether-lumefantrine and RDTs.
  Other Names: HFI
  Arms: Health Facility intervention
Other: Standard care — In the clusters randomized to standard care, standard care will include services typically provided by government-run facilities; we will not provide any additional support to these facilities. Health care will be provided to patients attending these facilities according to the usual standards; in-charges will continue to manage the facilities using their standard approach, no additional training will be provided to the health workers stationed at these facilities; and no support for staffing or supplies will be provided beyond what is supplied by the district and MoH.
  Arms: Standard of care

SUMMARY:
The investigators propose to assess whether an intervention to build capacity and improve delivery of drugs and diagnostics at government-run health facilities improves the health of children and quality of care delivered, as compared to 'standard care' currently available at health facilities, supplemented by services provided through the private sector and community-based interventions. The target population will be divided into 20 clusters, defined as the catchment area of lower-level public health facilities. Clusters will be randomized to the health facility intervention (HFI) or to standard care delivered from government-run health facilities, supplemented by services provided through the private sector and community-based interventions. The intervention is designed to address barriers to delivering quality care at health centers and will focus on three components: (1) training in-charges in health center management, (2) providing training to health workers in fever case management and patient-centered services, and (3) ensuring adequate supplies of artemether-lumefantrine and RDTs. Outcomes will be measured in three distinct populations: (1) cross-sectional surveys of children under 15 years randomly selected from households within the clusters; (2) a cohort of children under five randomly selected from households within the clusters and followed for 2 years; and (3) patients attending all government-run health facilities, including children under five and their caregivers participating in exit interviews on selected days every six months. The primary outcome of the study is prevalence of anemia in children under five.

DETAILED DESCRIPTION:
Study overview:

We are proposing to evaluate enhanced health facility-based care for malaria and febrile illnesses in children in Tororo district using a cluster randomized design. The health facility intervention (HFI) will aim to address barriers to achieving good quality health care that were identified in our formative research. The focus of our intervention will be providing RDTs and training health workers in management of both malaria and non-malarial febrile illnesses.

Study site:

The study will be conducted in Tororo district, an area with very high malaria transmission intensity. The estimated entomologic inoculation rate (EIR) in Tororo is 562 infective bites per person-year, and the prevalence of parasitemia among children aged 5-9 years is 63.5%. The five sub-counties of West Budama North Health Sub-district (Nagongera, Paya, Kirewa, Kisoko, and Petta), and two sub-counties of West Budama South Health Sub-district (Mulanda and Rubongi) will be included in the study population.

Study population:

Within the seven sub-counties, there are 22 lower-level government run health facilities, including 17 level II health centers (HC), and 5 level III HCs; 20 will be included in the randomization scheme.

Randomization:

The lower-level government-run health facilities in the study area will be the unit of randomization. Clusters will be defined as the catchment areas of the health centers, including households located within a 2km radius of the facilities. The clusters will be defined prior to randomization using the full census survey database. Households will be excluded from our sampling frame if they are > 2km from any health facility. The randomization will be conducted by an investigator who is not directly involved in the project. Health facilities will be stratified by level (HC IIs and HC IIIs). Because of the uneven numbers of HC IIs and IIIs, one of the HC IIIs without a laboratory will be 'demoted' and paired with a HC II to ensure even numbers. Restricted randomization will be employed to ensure balance on geographical location. Specifically, restrictions will be applied that exclude the allocation of all clusters originating from a single sub-county, or that are otherwise in close geographical proximity from being allocated to the same arm of the trial.

The Health Facility Intervention:

The intervention is designed to address barriers to delivering quality care at health centers and will focus on three components: (1) training in-charges in health center management, (2) providing training to health workers in fever case management and patient-centered services, and (3) ensuring adequate supplies of artemether-lumefantrine and RDTs.

1. Training in-charges:

   All in-charges of health centers randomized to the HFI will be trained in health center management. The purpose of this training is to equip in-charges with the skills and tools required to effectively and efficiently manage their health center. The training will include three components: (1) financial management, (2) supply management, and (3) information management.
2. Health worker training:

   A)Training in fever case management and use of RDTs All clinical staff will receive training in fever case management. Training will be based on the Integrated Malaria Management training package developed by the Joint Uganda Malaria Training Program (JUMP) team, and the RDT training guidelines which have been adopted and implemented by Uganda's MoH 'User's manual: Use of Rapid Diagnostic Tests (RDTs) for malaria in fever case management in Uganda'. The training program will be conducted by the JUMP training team over two weeks; the first two days will focus on theory, and will be followed by support supervision at the health facilities the next week. The training will be conducted in Tororo at a local health facility, and health workers will be trained in two small groups to ensure that work at the health facilities continues alongside the training. The impact of training on knowledge will be assessed using a pre-and post-training evaluation administered by the JUMP team. Additional support supervision will be conducted at 6 weeks and 6 months after the initial training and refresher training will be provided as needed.

   B)Training in patient-centered services The purpose of the Patient-Centered Services (PCS) training module is to identify and improve interpersonal interactions between health workers and patients. The module builds on the results of our formative research which identified several barriers to proving good quality health care at health facilities, including poor interpersonal interactions between health workers and community members resulting from poor communication skills, discriminatory behaviors of health workers, poor health worker motivation, and lack of patient-centered thinking. Through the PCS module, health workers will learn to recognize these challenges and develop skills for communicating and interacting with patients. The PCS module training will be implemented in a tiered approach to (1) all clinical staff, and (2) all health center support staff. All clinical staff, including in-charges, will receive the full PCS training package which includes self-observation tasks and specific emphasis on clinical and patient interaction challenges. Support staff including volunteers will receive a scaled-down PCS training package with specific emphasis on welcoming and guiding patients at the health facility. All training activities and workshops will be led by study personnel and trainers with experience in adult learning methodology.
3. Supply of AL and RDTs for malaria If the amount of AL provided to the intervention health centers by NMS is not adequate to meet demand, or if the procurement of AL fails, the project will supply supplemental AL. In addition, we will ensure adequate supplies of RDTs at all intervention health centers.

Evaluation procedures:

Outcomes will be measured in three distinct populations: (1) cross-sectional surveys of children under 15 years randomly selected from households within the clusters; (2) a cohort of children under five randomly selected from households within the clusters and followed for 2 years; and (3) patients attending all government-run health facilities, including children under five and their caregivers participating in exit interviews on selected days every six months.

1. Cross-sectional surveys will be conducted in randomly selected children under-five, and those between the ages of 5-15 years of age. The number of children sampled will be weighted according to the total population of each cluster to achieve a harmonic mean of 200 for each age category. A total of 8766 children will be sampled in each survey. Surveys will be conducted at baseline and then annually for each year; new populations of children will be selected for each survey. The survey will include a structured questionnaire administered to the primary caregiver, and a clinical and laboratory assessment of each child.
2. A Cohort of children under five will be enrolled from 25 households randomly selected from each cluster, for a total of 500 households. The cohort will be dynamic, in that all children within a household, who are under the age of five and who meet selection criteria, will be included. A household survey will be conducted at the start of the study. Children will undergo clinical and laboratory assessments at baseline and then every six months. Primary caregivers will be asked to prospectively collect information on the clinical symptoms of participating children and expenditures for health care using pictorial diaries. Study personnel will visit the households monthly to collect the diaries and administer a monthly questionnaire. Participants will be followed for approximately 18 months in total, the equivalent of approximately 12 months following roll-out of the intervention.
3. Patient Exit Interviews will be conducted with children under five and their caregivers at all health facilities. The purpose of the interviews is to evaluate for rational prescribing of ACTs, and to determine the level of satisfaction with the health facility visit. Three rounds of surveys are planned. In the first two surveys, 10 patients will be selected by convenience sampling from each facility to participate in the interviews (200 total per survey). In the final survey, 50 patients will be recruited to participate (1000 total in survey). In total, 1400 patients will participate in the interviews.

ELIGIBILITY:
FOR THE COHORT STUDY

Inclusion Criteria:

1. age < 5 years
2. agreement of parents or guardians to provide informed consent

Exclusion Criteria:

1) intention to move during the follow-up period

FOR THE CROSS-SECTIONAL SURVEY:

Inclusion Criteria:

1. age < 15 years
2. agreement of parents or guardians to provide informed consent
3. agreement of a child aged 8 years or older to provide assent.

Exclusion Criterion:

1) inability to locate the child.

Max Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25000 (Actual)
Dates: Start 2010-12; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of anemia in children under five in the cross-sectional surveys | annually
  Proportion of hemoglobin measurements < 11.0 g/dL as measured in cross sectional surveys. Anemia will be classified according to severity: mild (Hb 8.0 - 10.9), moderate (Hb 5.0 - 7.9), severe (Hb < 5.0).

SECONDARY OUTCOMES:
Prevalence of parasitemia in children under five in the cross-sectional surveys | annually
  Proportion of thick blood smears that are positive for asexual parasites
All-cause mortality | Annually
  Probability of dying between birth and five years of age, expressed per 1,000 live births
Incidence of hospitalizations in children under five in the cohort study | two years
  Overnight admission to a hospital or clinic
Incidence of illness episodes in children under five in the cohort study | Two years
  Episode of illness as reported by primary caregiver
Incidence of febrile episodes in children under five in the cohort study | Two years
  Episode of illness associated with fever as reported by primary caregiver
Prompt effective treatment of fever in children under five in the cohort study | Two years
  Proportion of children with fever treated within 24 hours of onset of symptoms with an ACT
Incidence of serious adverse events in children under five in the cohort study | Two years
  Any experience that results in death, life-threatening experience, hospitalization, persistent or significant disability or incapacity, or specific medical or surgical intervention to prevent one of the other serious outcomes
Prompt effective treatment of malaria in children under five in the cohort study | Two years
  Proportion of children with malaria (confirmed by a parasitological test) treated within 24 hours of onset of symptoms with an ACT
Appropriate treatment of malaria in children under five in the Patient Exit Interviews | Every six months
  Proportion of children under five with suspected malaria and a positive RDT result who are appropriately given an ACT + Proportion of children under five with suspected malaria and a negative RDT result who are not prescribed an ACT
Inappropriate treatment of malaria in children under five in the Patient Exit Interviews | Every six months
  Proportion of children under five with suspected malaria and a positive RDT result who are inappropriately given a non-ACT regimen
Patient satisfaction with health care in caregivers of children under five in the Patient Exit Interviews | Every six months
  Proportion of patients indicating they were satisfied with care provided at the health center in exit interviews
Patient attendance in the Health facility surveillance | Every two months
  Total number of patients attending health facilities and their characteristics, including age, sex,village of residence, and diagnosis
Stock-outs of ACTs in the Health facility surveillance | Every two months
  Days per month that AL supplied by NMS via the district is not available
Knowledge questionnaire scores for Health workers | Annually
  Proportion of questions answered correctly by clinicians following training in fever case management
Prevalence of anemia in children aged 5-15years in the cross-sectional surveys | annually
  Proportion of hemoglobin measurements < 11.0 g/dL as measured in cross sectional surveys. Anemia will be classified according to severity: mild (Hb 8.0 - 10.9), moderate (Hb 5.0 - 7.9), severe (Hb < 5.0).

OTHER OUTCOMES:
Antimalarial treatment incidence density for children under five in the cohort study | 2 years
  Number of antimalarial treatments given for treatment of fever/malaria over the period of follow-up
Inappropriate treatment of malaria in children under five in the Patient Exit Interviews | Every six months
  Proportion of children under five with suspected malaria and a negative RDT result who are inappropriately given an ACT + Proportion of children under five with suspected malaria and a positive RDT result who are not prescribed an ACT.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah G Staedke, MD, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Infectious Diseases Research Collaboration, Kampala, Uganda

REFERENCES:
- [Background] Staedke SG, Mwebaza N, Kamya MR, Clark TD, Dorsey G, Rosenthal PJ, Whitty CJ. Home management of malaria with artemether-lumefantrine compared with standard care in urban Ugandan children: a randomised controlled trial. Lancet. 2009 May 9;373(9675):1623-31. doi: 10.1016/S0140-6736(09)60328-7. Epub 2009 Apr 9. PMID 19362361
- [Background] Hopkins H, Talisuna A, Whitty CJ, Staedke SG. Impact of home-based management of malaria on health outcomes in Africa: a systematic review of the evidence. Malar J. 2007 Oct 8;6:134. doi: 10.1186/1475-2875-6-134. PMID 17922916
- [Derived] Chandler CI, DiLiberto D, Nayiga S, Taaka L, Nabirye C, Kayendeke M, Hutchinson E, Kizito J, Maiteki-Sebuguzi C, Kamya MR, Staedke SG. The PROCESS study: a protocol to evaluate the implementation, mechanisms of effect and context of an intervention to enhance public health centres in Tororo, Uganda. Implement Sci. 2013 Sep 30;8:113. doi: 10.1186/1748-5908-8-113. PMID 24079992
- [Derived] Staedke SG, Chandler CI, DiLiberto D, Maiteki-Sebuguzi C, Nankya F, Webb E, Dorsey G, Kamya MR. The PRIME trial protocol: evaluating the impact of an intervention implemented in public health centres on management of malaria and health outcomes of children using a cluster-randomised design in Tororo, Uganda. Implement Sci. 2013 Sep 30;8:114. doi: 10.1186/1748-5908-8-114. PMID 24079295
- See also: Infectious Diseases Research Collaboration (UMSP, MU-UCSF) — http://www.muucsf.org